CLINICAL TRIAL: NCT03288948
Title: Binocular Amblyopia Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eileen Birch, Senior Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062010-105; R01EY022313 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Contrast Increment (Active Comparator)
  Interventions: Other: Binocular games for treatment of amblyopia
- Reduced Contrast Increment (Experimental)
  Interventions: Other: Binocular games for treatment of amblyopia
- No Contrast Increment (Experimental)
  Interventions: Other: Binocular games for treatment of amblyopia

INTERVENTIONS:
Other: Binocular games for treatment of amblyopia — playing binocular games on a tablet platform 1 hour per day 5 days per week with reduced contrast for the fellow eye and high contrast for the amblyopic eye

SUMMARY:
To evaluate the effectiveness of enhanced binocular amblyopia treatments in achieving a more complete and stable recovery.

DETAILED DESCRIPTION:
To date, all studies of contrast-rebalanced binocular amblyopia treatment games used the same 10% per day contrast-increment that was designed for short-term intervention studies lasting 1-4 weeks; i.e., after 18 days of successful game play, both eyes viewed 100% contrast (no contrast-rebalancing).This study will investigate two alternative protocols designed to extend the game treatment period beyond 4 weeks to allow for more complete recovery of visual acuity. The new protocols will be compared with the original 10% contrast-increment game protocol in an 8-week 3-arm RCT to determine whether one or both of the new protocols is more effective than the current 10% increment.

Based on pilot data, we expect about 40% of amblyopic children to achieve normal visual acuity in 8 weeks. In an effort to also promote recovery of binocular vision, children who attain ≤0.4 logMAR at 8 weeks will be enrolled in stereoacuity training at the 8-week visit for the next 4 weeks. Children with residual amblyopia (BCVA >0.4 logMAR) at the 8-week visit will be provided with dichoptic movies for additional amblyopia treatment for another 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 4-10 y
* male and female
* strabismic, anisometropic, or combined mechanism amblyopia
* amblyopic eye best-corrected visual acuity 0.3-0.8 logMAR
* fellow eye best-corrected visual acuity ≤0.1 logMAR
* interocular visual acuity difference ≥0.3 logMAR
* wearing glasses (if needed) for 8 weeks or no change visual acuity with glasses at 2 visits

  * 4 weeks apart.
* child's ophthalmologist and family must be willing to forgo patching treatment during the 12-week study period
* parent's informed consent
* child must demonstrate understanding and ability to play binocular games

Exclusion Criteria:

* prematurity ≥8 weeks
* coexisting ocular or systemic disease
* developmental delay
* strabismus >5pd
* any binocular amblyopia treatment in the past 3 months

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity of the amblyopic eye | baseline vs 8 weeks
  ATS-HOTV for age 4-6.9 years or E-ETDRS for age 7-10.9 years

SECONDARY OUTCOMES:
Change in visual acuity of the amblyopic eye | baseline vs 2, 4, 6, and 12 weeks
  ATS-HOTV for age 4-6.9 years or E-ETDRS for age 7-10.9 years
Change in stereoacuity | baseline vs 2, 4, 6, 8, 12 weeks
  Randot Preschool Stereoacuity Test
Change in suppression | baseline vs 2, 4, 6, 8, 12 weeks
  Dichoptic Letter Chart

OTHER OUTCOMES:
Change in accommodation | baseline vs 8 week
  Accuracy of accommodation to a near target (Grand Seiko)
Change in motion perception | baseline vs 8 weeks
  Motion-defined form
Change in fixation stability | baseline vs 8 weeks
  Bivariate contour ellipse area
Reading speed | baseline vs 4 and 8 weeks
  Reading speed in wpm
Fine motor skills | baseline vs 4 and 8 weeks
  M-ABC
Self-perception | baseline vs 8 weeks
  self-perception questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
we will only share aggregated data

REFERENCES:
- [Derived] Jost RM, Kelly KR, Birch EE. Risk of recurrence after cessation of dichoptic, binocular treatment of amblyopia. J AAPOS. 2023 Oct;27(5):298-300. doi: 10.1016/j.jaapos.2023.06.009. Epub 2023 Aug 23. PMID 37619861
- [Derived] Jost RM, Kelly KR, Hunter JS, Stager DR Jr, Luu B, Leffler JN, Dao L, Beauchamp CL, Birch EE. A randomized clinical trial of contrast increment protocols for binocular amblyopia treatment. J AAPOS. 2020 Oct;24(5):282.e1-282.e7. doi: 10.1016/j.jaapos.2020.06.009. Epub 2020 Oct 9. PMID 33045374